CLINICAL TRIAL: NCT06951347
Title: Impact of Prophylactic Sodium Supplementation on Hospital Outcomes in Infants and Children With Pneumonia. A Randomized Controlled Trial
Brief Title: Prophylactic Sodium Supplementation for Children Hospitalized With Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Organization for Teaching Hospitals and Institutes (Other)
Responsible Party: Principal Investigator, Marwa Taha, MD, Fellow of Pediatrics, Mataria Teaching Hospital (Principal Investigator), General Organization for Teaching Hospitals and Institutes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HM000174
Record Dates: First submitted 2025-04-19; First posted 2025-04-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Childhood Pneumonia
MeSH Terms: interventions — World Health Organization oral rehydration solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Dietary Supplement: Oral Rehydration Solution
- Control Group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Oral Rehydration Solution — one sachet every day for 3 days
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to study the impact of sodium supplementation on hospital outcomes of children with pneumonia.

It aims to answer:

* Does sodium supplementation lower the length of hospital stay in children with pneumonia?
* Does potassium supplementation lower the length of hospital stay in children with pneumonia?

Researchers will compare the intervention arm to the control arm to see if the intervention lowers the length of hospital stay.

Participants will:

• Take one sachet of oral rehydration solution (ORS) every day for 3 days.

DETAILED DESCRIPTION:
The study is a randomized clinical trial that will be conducted on hospitalized children with pneumonia after considering exclusion criteria.

The enrolled children will be randomly divided into two groups: the intervention group and the control group. The intervention group will receive the ORS daily for 3 days.

All children will be followed until discharge from the hospital, and their clinical outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children aged between 1 month and 5 years.
* Patients diagnosed with pneumonia according to World Health Organization (WHO) criteria.

Exclusion Criteria:

* Children with other comorbidities.
* Those whose parents will show disapproval for the participation of the study.
* Children on medications that affect sodium and potassium levels.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
The difference in hospital length of stay between hospitalized children with pneumonia who received oral rehydration solution and those who did not receive it | Children will be followed until discharge from the hospital, an average of one week.
  Evaluation of effect of oral rehydration solution supplementation by assessing the length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Taha, MD, Principal Investigator — Mataria Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Cairo, Egypt; Hoda Atef Abdelsattar Ibrahim, MD, Principal Investigator — Faculty of Medicine, Cairo University, Cairo, Egypt
Locations (1):
- Mataria Teaching Hospital, Cairo, Egypt